CLINICAL TRIAL: NCT04703998
Title: Arthroscopic Rotator Cuff Repair Augmented With Platelet Rich Plasma. Prospective Randomized Controlled Trial.
Brief Title: Arthroscopic Rotator Cuff Repair Augmented With Platelet Rich Plasma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Italiano de Buenos Aires (Other)
Responsible Party: Principal Investigator, LUCIANO ANDRES ROSSI, Pincipal investigator, Hospital Italiano de Buenos Aires
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5702
Record Dates: First submitted 2021-01-03; First posted 2021-01-11 (Actual); Last update posted 2022-12-22 (Actual); Status verified 2022-12

CONDITIONS: Rotator Cuff Tears
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arthroscopic rotator cuff repair and platelet rich plasma (Experimental): A standard double-row arthroscopic rotator cuff repair will be performed and at the end of the procedure 10 ml of autologous platelet-rich plasma will be placed under direct vision at the tendon-bone interface.
  Interventions: Procedure: Arthroscopic rotator cuff repair; Biological: platelet rich plasma
- Arthroscopic rotator cuff repair (Active Comparator): A standard double-row arthroscopic rotator cuff repair will be performed.
  Interventions: Procedure: Arthroscopic rotator cuff repair

INTERVENTIONS:
Procedure: Arthroscopic rotator cuff repair — A double-row rotator cuff repair will be performed.
Biological: platelet rich plasma — A single dose of 10 ml of autologous platelet rich plasma at the bone-tendon interfase will be administered.
  Arms: Arthroscopic rotator cuff repair and platelet rich plasma

SUMMARY:
Purpose: To assess whether the use of platelet-rich plasma used as an adjuvant to arthroscopic rotator cuff repairs modify the rate of re-tears (measured by MRI) compared to a control group that only underwent the isolated arthroscopic repair. Hypothesis: Platelet rich plasma used as an adjuvant to arthroscopic rotator cuff repairs decrease the rate of retears.

DETAILED DESCRIPTION:
Platelet-rich plasma used as an adjuvant to arthroscopic rotator cuff repairs modify the rate of re-tears (measured by MRI) compared to a control group that only underwent the isolated arthroscopic repair.

ELIGIBILITY:
Inclusion Criteria:

* Adults between 50 and 75 years with a defined complete rotator cuff tear as compatible clinical and confirmation by magnetic resonance imaging (MRI).
* Minimum of 3 months of failed conservative treatment (anti-inflammatory, physical therapy and infiltration with corticosteroids)

Exclusion Criteria:

* Refusal to participate or informed consent,
* Revision surgery,
* Partial repair,
* Patients with shoulder osteoarthritis> 2
* Advanced fat infiltration of the rotator cuff muscles (STAGE 3 or 4)
* Systemic or rheumatoid arthritis,
* Uncontrolled diabetes, (patients for whom surgery is contraindicated in the preoperative evaluation by the clinician and anesthesiologist)
* Acute or chronic infections of the shoulder to be operated on
* Ongoing cancer chemotherapy therapies
* Sepsis, septic arthritis, osteomyelitis or other ongoing infectious processes;
* Previous operations on the affected shoulder,
* Patients with autoimmune diseases;
* Pregnant

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2021-01-03 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Comparison of re-tear rates between groups. | 6 months
  Postoperative MRI to assess the structural integrity of the repaired rotator cuff.

SECONDARY OUTCOMES:
Change From baseline in shoulder functional scores at 3, 6 and 12 months | baseline, 3, 6, and 12 months
  The ASES score (American Shoulder and Elbow Surgeons) and the Constant score will be used. Both scores assess the general function of the shoulder in different activities of daily life, global mobility of the shoulder and pain with usual tasks. They are scores ranging from 0 to 100. Both scores are validated and are the reference scores for clinical research on rotator cuff pathology
Change From baseline in pain at 3, 6 and 12 months | baseline, 3, 6, and 12 months
  The visual analog scale (VAS) will be used to assess the level of pain during activities of daily living. 0 will be considered as "no pain" and 10 as "the worst pain of his life."
Number of Participants With Treatment-Related Adverse Events | 3, 6, and 12 months
  Adverse effects and postoperative complications will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Luciano Rossi, MD, Principal Investigator — Hospital Italiano de Buenos Aires
Locations (1):
- Hospital Italiano de Buenos Aires, CABA, Argentina

IPD SHARING:
Plan to Share IPD: Yes
We are planning on sharing the study protocol and the tables contaning all outcomes for every individual patient
Supporting Information: Study Protocol, CSR
Time Frame: 2 years
Access Criteria: The IPD may be requested to the principal investigator contacting him through e-mail at luciano.rossi@hospitalitaliano.org.ar

REFERENCES:
- [Derived] Rossi LA, Gorodischer TD, Camino P, Brandariz RN, Tanoira I, Piuzzi NS, Ranalletta M. Leukocyte-Poor Platelet-Rich Plasma as an Adjuvant to Arthroscopic Rotator Cuff Repair Reduces the Retear Rate But Does Not Improve Functional Outcomes: A Double-Blind Randomized Controlled Trial. Am J Sports Med. 2024 May;52(6):1403-1410. doi: 10.1177/03635465241239062. Epub 2024 Apr 8. PMID 38587033